CLINICAL TRIAL: NCT04702009
Title: Efficacy and Safety of First-line Anti-PD-1/PD-L1 Monoclonal Antibody in Combination With Chemotherapy vs. Anti-PD-1/PD-L1 Monoclonal Antibody, Chemotherapy, in Combination With Bronchoscopy-assisted Interventional Therapy in the Treatment of Patients With Advanced Central Non-small Cell Lung Cancer, a Randomized Controlled, Prospective Clinical Trial
Brief Title: Efficacy and Safety of First-line Anti-PD-1/PD-L1 Monoclonal Antibody in Combination With Chemotherapy and Bronchoscopy-assisted Interventional Therapy in Patients With Advanced Central Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Yayi He, Associate Chief Physician, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021HY017
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Advanced Lung Carcinoma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-PD-1/PD-L1 Monoclonal Antibody in Combination With Chemotherapy (Active Comparator): Anti-PD-1/PD-L1 Monoclonal Antibody in Combination With Chemotherapy
  Interventions: Drug: Anti-PD-1/PD-L1 Monoclonal Antibody，Chemotherapy
- Anti-PD-1/PD-L1 Antibody, Chemotherapy, and Bronchoscopy-assisted Interventional Therapy (Experimental): Anti-PD-1/PD-L1 Antibody, Chemotherapy, and Bronchoscopy-assisted Interventional Therapy
  Interventions: Drug: Anti-PD-1/PD-L1 Monoclonal Antibody，Chemotherapy; Device: Bronchoscopy-assisted Interventional Therapy

INTERVENTIONS:
Drug: Anti-PD-1/PD-L1 Monoclonal Antibody，Chemotherapy — Anti-PD-1/PD-L1 monoclonal antibody (approved anti-PD-1/PD-L1 monoclonal antibody)；albumin paclitaxel/docetaxel + carboplatin (albumin paclitaxel 130mg/m2, d1 d8, Docetaxel 75mg/m2, carboplatin AUC=5, d1, every 21 days, 4 cycles of chemotherapy; immunotherapy no more than 2 years)
Device: Bronchoscopy-assisted Interventional Therapy — Bronchoscopy-assisted interventional therapy (1 time before chemotherapy or 2 times before chemotherapy and before the third cycle of treatment)
  Arms: Anti-PD-1/PD-L1 Antibody, Chemotherapy, and Bronchoscopy-assisted Interventional Therapy

SUMMARY:
Lung cancer is one of the malignant tumors with high morbidity and mortality. Several PD-1/PD-L1 immune checkpoint inhibitors have been approved for the treatment of advanced non-small cell lung cancer (NSCLC). However, its overall effective population is only 20%, and even in studies of enriched populations (such as PD-L1 ≥ 50%), its single-drug effective rate is only about 40%. Therefore, this study aims to explore the efficacy and safety of anti-PD-1/PD-L1 monoclonal antibodies and chemotherapy in combination with bronchoscopy-assisted lnterventional therapy in the first-line treatment of advanced central non-small cell lung cancer. We conducted a randomized controlled, prospective clinical trial to examine the efficacy, safety, and mechanism of anti-PD-1/PD-L1 monoclonal antibodies, chemotherapy, in combination with bronchoscopy-assisted interventional therapy vs anti-PD-1/PD-L1 monoclonal antibody in combination with chemotherapy as the first-line treatment of patients with advanced central NSCLC.

DETAILED DESCRIPTION:
Lung cancer is one of the malignant tumors with high morbidity and mortality. Most patients with lung cancers are already in advanced stages when diagnosed, and the 5-year survival rate of advanced lung cancer is less than 5%. Therefore, exploring effective treatments is of great significance for improving the survival and quality of life of patients with lung cancer. Immunotherapy represented by immune checkpoint inhibitors has received widespread attention in the field of lung cancer, and several PD-1/PD-L1 immune checkpoint inhibitors have been approved for the treatment of advanced non-small cell lung cancer (NSCLC).However, its overall effective population is only 20%, even in studies of enriched populations (such as PD-L1 ≥ 50%), its single-drug effective rate is only about 40%. Therefore, this study aims to explore the efficacy and safety of anti-PD-1/PD-L1 monoclonal antibodies and chemotherapy in combination with bronchoscopy-assisted interventional therapy in the first-line treatment of advanced central non-small cell lung cancer. We conducted a randomized controlled, prospective clinical trial to examine the efficacy, safety and mechanism of anti-PD-1/PD-L1 monoclonal antibodies and chemotherapy in combination with bronchoscopy-assisted interventional therapy versus anti-PD-1/PD-L1 monoclonal antibody in combination with chemotherapy as the first-line treatment of patients with advanced central NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1) Patients volunteer to participate in clinical studies and sign an informed consent (ICF), and are willing to follow and able to complete all trial procedures.

2)18-75 years of age 3) All patients included are diagnosed with lung cancer detected by fibrous bronchoscope or percutaneous lung puncture biopsy, and are confirmed as NSCLC by Immunohistochemistry.

4) Obstruction-type central lung cancer that cannot be surgically removed. 5) Patients without EGFR, ALK, and ROS mutation. 6) Patients have not previously received systemic treatment for phase IV NSCLC or patients receiving the adjuvant or neoadjuvant therapy for more than 6 months before the diagnosis of phase IV NSCLC.

7) Within 4 weeks, at least one measurable lesions are required for researchers to evaluate in accordance with RECIST 1.1 requirements.

8) Appropriate tumor tissues for PD-L1 expression level determination are required.

9) Relevant laboratory tests indicate tolerance for chemotherapy, immunotherapy, and bronchoscopy.

Exclusion Criteria:

1. Patients with uncertain diagnosis.
2. Non-central NSCLC patients.
3. Patients with contraindications to chemotherapy or immunotherapy.
4. Bronchoscopy is contraindicated in patients.
5. Patients have other active malignancies. Patients with cured limited tumors, such as skin substrate cell carcinoma, skin squamous cancer, superficial bladder cancer, carcinoma in situ of prostate, carcinoma in situ of cervix, and breast in-place cancer, can be included.
6. Patients with human immunodeficiency virus (HIV) infection.
7. Patients with infection of active tuberculosis.
8. Patients have received a live vaccines within 28 days of the first drug use. Patients receiving inactivated viral vaccines to treat seasonal influenza are allowed, but inactivated live influenza vaccines with intracn nasal drugs are not allowed.
9. Pregnant or lactating women.
10. Patients have a known history of psychosophedic substance abuse or drug abuse;
11. The researchers determined that there may be other factors that might have contributed to the early termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-20 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 6 weeks
  To evaluate the objective response rate (ORR) in the first-line treatment of patients with advanced central NSCLC

SECONDARY OUTCOMES:
disease control rate (DCR) | 6 weeks
  To evaluate the disease control rate (DCR) in the first-line treatment of patients with advanced central NSCLC
progression free survival (PFS) | 1 year
  To evaluate the progression free survival (PFS) in the first-line treatment of patients with advanced central NSCLC
overall survival (OS) | 2 years
  To evaluate the overall survival (OS) in the first-line treatment of patients with advanced central NSCLC
Number of participants with treatment-related adverse events (AE) as assessed by CTCAE v4.0 | 2 years
  To evaluate the side effects in the first-line treatment of patients with advanced central NSCLC
quality of life (QoL) | 2 years
  To evaluate the quality of life (QoL) in the first-line treatment of patients with advanced central NSCLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] He Y, Rozeboom L, Rivard CJ, Ellison K, Dziadziuszko R, Yu H, Zhou C, Hirsch FR. MHC class II expression in lung cancer. Lung Cancer. 2017 Oct;112:75-80. doi: 10.1016/j.lungcan.2017.07.030. Epub 2017 Jul 29. PMID 29191604
- [Background] He Y, Rozeboom L, Rivard CJ, Ellison K, Dziadziuszko R, Yu H, Zhou C, Hirsch FR. PD-1, PD-L1 Protein Expression in Non-Small Cell Lung Cancer and Their Relationship with Tumor-Infiltrating Lymphocytes. Med Sci Monit. 2017 Mar 9;23:1208-1216. doi: 10.12659/msm.899909. PMID 28275222
- [Background] Deng J, Zhao S, Zhang X, Jia K, Wang H, Zhou C, He Y. OX40 (CD134) and OX40 ligand, important immune checkpoints in cancer. Onco Targets Ther. 2019 Sep 6;12:7347-7353. doi: 10.2147/OTT.S214211. eCollection 2019. PMID 31564917
- [Background] He Y, Yu H, Rozeboom L, Rivard CJ, Ellison K, Dziadziuszko R, Suda K, Ren S, Wu C, Hou L, Zhou C, Hirsch FR. LAG-3 Protein Expression in Non-Small Cell Lung Cancer and Its Relationship with PD-1/PD-L1 and Tumor-Infiltrating Lymphocytes. J Thorac Oncol. 2017 May;12(5):814-823. doi: 10.1016/j.jtho.2017.01.019. Epub 2017 Jan 26. PMID 28132868
- [Background] He Y, Jia K, Dziadziuszko R, Zhao S, Zhang X, Deng J, Wang H, Hirsch FR, Zhou C. Galectin-9 in non-small cell lung cancer. Lung Cancer. 2019 Oct;136:80-85. doi: 10.1016/j.lungcan.2019.08.014. Epub 2019 Aug 16. PMID 31454748